CLINICAL TRIAL: NCT04840745
Title: A Randomized, Single-blinded, Parallel Design Phase I Clinical Trial to Investigate the Safety and Pharmacokinetics/Pharmacodynamics of CKD-841 A-1, CKD-841 D or Leuplin Inj. After Subcutaneous Injection in Postmenopausal Female
Brief Title: The Safety and Pharmacokinetic/Pharmacodynamic Study of CKD-841 in Postmenopausal Female, Phase 1
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Collaborators: Severance Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: A55_03PK2023
Record Dates: First submitted 2021-04-08; First posted 2021-04-12 (Actual); Last update posted 2021-04-19 (Actual); Status verified 2021-04

CONDITIONS: Early Puberty
Keywords: CKD-841; Postmenopausal; Leuplin
MeSH Terms: conditions — Puberty, Precocious

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- CKD-841 A-1(=leuprorelin acetate 3.75mg) (Experimental): Investigational drug(=CKD-841 A-1) is prescribed single injection dose by subcutaneous to 8 of randomized subjects once.
  Interventions: Drug: CKD-841 A-1 3.75mg
- CKD-841 A-1(=leuprorelin acetate 1.88mg) (Experimental): Investigational drug(=CKD-841 A-1) is prescribed single injection dose by subcutaneous to 8 of randomized subjects once.
  Interventions: Drug: CKD-841 A-1 1.88mg
- CKD-841 D(=leuprorelin acetate 2.92mg) (Experimental): Investigational drug(=CKD-841 D) is prescribed single injection dose by subcutaneous to 8 of randomized subjects once.
  Interventions: Drug: CKD-841 D 2.92mg
- Leuplin Inj.(=leuprorelin acetate 3.75mg) (Active Comparator): Investigational drug(=Leuplin Inj.)is prescribed single injection dose by subcutaneous to 8 of randomized subjects once.
  Interventions: Drug: Leuplin Inj. 3.75 mg

INTERVENTIONS:
Drug: CKD-841 A-1 3.75mg — Single injection, subcutaneous injection
  Other Names: CKD-841
  Arms: CKD-841 A-1(=leuprorelin acetate 3.75mg)
Drug: CKD-841 A-1 1.88mg — Single injection, subcutaneous injection
  Other Names: CKD-841
  Arms: CKD-841 A-1(=leuprorelin acetate 1.88mg)
Drug: CKD-841 D 2.92mg — Single injection, subcutaneous injection
  Other Names: CKD-841
  Arms: CKD-841 D(=leuprorelin acetate 2.92mg)
Drug: Leuplin Inj. 3.75 mg — Single injection, subcutaneous injection
  Other Names: Leuplin.Inj
  Arms: Leuplin Inj.(=leuprorelin acetate 3.75mg)

SUMMARY:
A randomized, single-blinded, parallel design phase I clinical trial to investigate the safety and pharmacokinetics/pharmacodynamics of CKD-841 A-1, CKD-841 D or Leuplin Inj. after subcutaneous injection in postmenopausal female

DETAILED DESCRIPTION:
To investigate the safety and pharmacokinetics/pharmacodynamics of CKD-841 A-1, CKD-841 D or Leuplin Inj. 3.75 mg after subcutaneous injection in postmenopausal female

ELIGIBILITY:
Inclusion Criteria:

* Healthy menopausal female
* β-hCG is negative at screening and before administration of investigational drug
* Infertility by sterilization operation before 5 months from screening excluding ovarian cancer, uterine cancer etc.
* Bwt ≥ 50Kg and Body Mass Index (BMI) ≥ 18.5 and < 28.0

Exclusion Criteria:

* History or current condition of disease related to Hepato-biliary system, renal system, nervous system, mental illness, immune system, respiratory system, endocrine system, hemato-oncology, circulatory system, musculoskeletal system or except for that, significant clinical disease
* Uncontrolled diabetes mellitus in the last three months
* Pregnancy or breast feeding
* History of taking medicine such as Leuprorelin acetate or similar affiliation drug within 12 weeks before administration of investigational drug
* Has hypersensitivity to the active ingredient or excipients or same affiliation drug of the investigational drug, hypersensitivity of a medicine contained gelatin especially

Min Age: 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2021-04 (Estimated); Primary Completion 2021-10 (Estimated); Study Completion 2021-11 (Estimated)

PRIMARY OUTCOMES:
PK(Cmax) | From before injection to up to 1008 hours post injection
  Cmax(Maximum concentration of drug in plasma) of Leuprorelin
PK(AUClast) | From before injection to up to 1008 hours post injection
  AUClast(Area under the plasma drug concentration-time curve to last measurement) of Leuprorelin
PK(AUCinf) | From before injection to up to 1008 hours post injection
  AUCinf(Area under the plasma drug concentration-time curve extrapolated to infinity) of Leuprorelin
PK(AUC7-t) | From before injection to up to 1008 hours post injection
  AUC7-t(Area under the plasma drug concentration-time curve from 7 days to last measurement) of Leuprorelin
PK(CL/F) | From before injection to up to 1008 hours post injection
  CL/F(Apparent Clearance) of Leuprorelin
PK(Vd/F) | From before injection to up to 1008 hours post injection
  Vd/F(Apparent Volume of Distribution) of Leuprorelin
PK(Tmax) | From before injection to up to 1008 hours post injection
  Tmax(Time to Cmax/Time to Emax) of Leuprorelin
PK(t1/2) | From before injection to up to 1008 hours post injection
  t1/2(Terminal elimination half-life) of Leuprorelin
PD(AUEC0-42d below baseline) | From before injection to up to 1008 hours post injection
  AUEC0-42d below baseline((AUEC that is below the baseline from 0 h to 42 days)) of the rate of change(%) relative to the base of the LH (Luteinizing Hormone), FSH (Follicular Stimulating Hormone), and Estradiol respectively.
PD(AUEC0-28d below baseline) | From before injection to up to 1008 hours post injection
  AUEC0-28d below baseline(AUEC that is below the baseline from 0 h to 28 days) of the rate of change(%) relative to the base of the LH (Luteinizing Hormone), FSH (Follicular Stimulating Hormone), and Estradiol respectively.
PD(Area under the response (% change from baseline) curve) | From before injection to up to 1008 hours post injection
  AUEC(Area under the response (% change from baseline) curve) above baseline of the rate of change(%) relative to the base of the LH (Luteinizing Hormone), FSH (Follicular Stimulating Hormone), and Estradiol respectively.
PD(Tmax) | From before injection to up to 1008 hours post injection
  Tmax(Time to Cmax/Time to Emax) of the rate of change(%) relative to the base of the LH (Luteinizing Hormone), FSH (Follicular Stimulating Hormone), and Estradiol respectively.
PD(Tmin) | From before injection to up to 1008 hours post injection
  Tmin(Time to Emin) of the rate of change(%) relative to the base of the LH (Luteinizing Hormone), FSH (Follicular Stimulating Hormone), and Estradiol respectively.
PD(Emax) | From before injection to up to 1008 hours post injection
  Emax(Maximum % change from baseline of LH/FSH/Estradiol) of the rate of change(%) relative to the base of the LH (Luteinizing Hormone), FSH (Follicular Stimulating Hormone), and Estradiol respectively.
PD(Emin) | From before injection to up to 1008 hours post injection
  Emin(Minimum % change from baseline of LH/FSH/Estradiol) of the rate of change(%) relative to the base of the LH (Luteinizing Hormone), FSH (Follicular Stimulating Hormone), and Estradiol respectively.

SECONDARY OUTCOMES:
Safety Assessment by evaluating adverse events(AEs). | From day1 to day 56
  Assessment of the safety of subjects by evaluating adverse events(AEs).

CONTACTS AND LOCATIONS:
Overall Officials: Min Soo Park, Ph.D, Principal Investigator — Severance Hospital
Locations (1):
- Severance Hospital, Seoul, Yonsei-ro, Seodaemun-gu 50-1, South Korea

IPD SHARING:
Plan to Share IPD: No